CLINICAL TRIAL: NCT01630980
Title: Effect of Tree Nuts on Glycemic Control and Features of the Metabolic Syndrome: A Systematic Review and Meta-analysis of Controlled Dietary Trials to Provide Evidence-based Guidance for Nutrition Guidelines Development
Brief Title: Meta-analyses of the Effect of Tree Nuts on Glycemic Control and Features of the Metabolic Syndrome
Status: Completed | Type: Observational
Sponsor: John Sievenpiper (Other)
Collaborators: The International Tree Nut Council Nutrition Research & Education Foundation (Unknown); Canada Research Chairs Endowment of the Federal Government of Canada (Other Government); Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Sponsor-Investigator, John Sievenpiper, Knowledge Synthesis Lead, University of Toronto
Organization: University of Toronto (Other)
Other Study IDs: INC 2012 KRS
Record Dates: First submitted 2012-05-18; First posted 2012-06-28 (Estimated); Last update posted 2015-05-27 (Estimated); Status verified 2015-05

CONDITIONS: Diabetes; Prediabetes; Dysglycemia; Overweight; Obesity; Dyslipidemia; Hypertension; Metabolic Syndrome; Cardiovascular Diseases
Keywords: Systematic review and meta-analysis; Evidence-based medicine (EBM); Evidence-based nutrition (EBN); Clinical practice guidelines; Clinical trials; Tree nuts; Cardiometabolic risk factors; Triglycerides; Cholesterol; Glycemic control; Insulin resistance; Body weight; Blood pressure
MeSH Terms: conditions — Diabetes Mellitus; Prediabetic State; Overweight; Obesity; Dyslipidemias; Hypertension; Metabolic Syndrome; Cardiovascular Diseases; Insulin Resistance; Body Weight

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Tree nuts — Almonds, Brazil nuts, cashews, hazelnuts, macadamia nuts, pecans, pine nuts, pistachios and walnuts in whole, meal, or flour form

SUMMARY:
Tree nuts (almonds, Brazil nuts, cashews, hazelnuts, macadamia nuts, pecans, pine nuts, pistachios and walnuts) are an important source of unsaturated fatty acids, vegetable protein, and fibre, as well as minerals, vitamins, and phytonutrients. Although heart disease risk reduction claims for nuts have been permitted in the U.S. and general dietary guidelines and recommendations from heart associations recommend the consumption of nuts for heart protection, diabetes associations have not addressed nuts in their most recent recommendations. This omission is despite heart disease being a major cause of death in diabetes. There remains insufficient information on the usefulness of these foods in diabetes. To improve evidence-based guidance for tree nut recommendations, the investigators propose to conduct a systematic review of the effect of tree nuts on diabetes control and features of the metabolic syndrome. The systematic review process allows the combining of the results from many small studies in order to arrive at a pooled estimate, similar to a weighted average, of the true effect. The investigators will be able to explore whether eating tree nuts has different effects between men and women, in different age groups and background disease states, and whether or not the effect of tree nuts depends on the dose and background diet. The findings of this proposed knowledge synthesis will help improve the health of Canadians through informing diabetes association recommendations and heart association recommendations where they relate to diabetes.

DETAILED DESCRIPTION:
Background: Tree nuts (almonds, Brazil nuts, cashews, hazelnuts, macadamia nuts, pecans, pine nuts, pistachios and walnuts)are an important source of unsaturated fatty acids, vegetable protein, and fibre, as well as minerals, vitamins, and phytonutrients. Although the dietary guidelines for Americans and American Heart Association (AHA) recommend the consumption of nuts for cardiovascular risk reduction and the US Food and Drug Administration (FDA) issued a qualified coronary heart disease (CHD) risk reduction claim for nuts, none of the diabetes associations have addressed nuts in their most recent recommendations. This omission is despite CHD being a major cause of death in diabetes. Several trials have been undertaken in diabetes, some of which, including the largest to date by our group, have demonstrated advantages in glycemic control. Although the remaining trials have failed to show a significant improvement in glycemic control, the direction of the effect has favored nuts, along with improvements in complementary markers of metabolic control.

Need for a review: The lack of high quality data in this area to support diabetes recommendations represents an urgent call for stronger evidence. A systematic review and meta-analysis of controlled feeding trials remains the "Gold Standard" of evidence for nutrition guidelines development.

Objective: To provide evidence-based guidance for diabetes guidelines, we will conduct two systematic reviews and meta-analyses of controlled feeding trials to assess the effect of tree nuts (almonds, Brazil nuts, cashews, hazelnuts, macadamia nuts, pecans, pine nuts, pistachios and walnuts) on cardiometabolic control: (1) "Tree nuts and glycemic control" and (2) "Tree nuts and features of the metabolic syndrome".

Design: The planning and conduct of the proposed meta-analyses will follow the Cochrane handbook for systematic reviews of interventions. The reporting will follow the Preferred Reporting Items for Systematic reviews and Meta-Analyses (PRISMA) guidelines.

Data sources: MEDLINE, EMBASE, CINAHL and The Cochrane Central Register of Controlled Trials will be searched using appropriate search terms.

Study selection: Intervention trials that investigate the effect of exchanging nuts for other diets on cardiometabolic risk outcomes in humans will be included. Studies that are <3-weeks diet duration, lack a control, or report non-isocaloric comparisons will be excluded.

Data extraction: Independent investigators (≥2) will extract information about study design, sample size, subject characteristics, nut form, dose, follow-up, and the composition of the background diets. Mean±SEM values will be extracted for all endpoints. Standard computations and imputations will be used to derive missing variance data. Risk of bias and study quality will be assessed using the risk of bias tool and the Heyland Methodological Quality Score (MQS), respectively.

Outcomes: The two proposed analyses will assess a set of outcomes related to a different area of cardiometabolic control: (1) glycemic control (glycated blood proteins[HbA1c, fructosamine, glycated albumin], fasting glucose, fasting insulin, and the homeostasis model assessment of insulin resistance [HOMA-IR]) and (2) harmonized metabolic syndrome features (waist circumference, TG, HDL-C, blood pressure, fasting glucose).

Data synthesis: Pooled analyses will be conducted using the Generic Inverse Variance method with random effects models. Random-effects models will be used even in the absence of statistically significant between-study heterogeneity, as they yield more conservative summary effect estimates in the presence of residual heterogeneity. Exceptions will be made for the use of fixed-effects models where there is <5 included trials irrespective of heterogeneity or small trials are being pooled with larger more precise trials in the absence of statistically significant heterogeneity. Paired analyses will be applied to all crossover trials. Heterogeneity will be tested by Cochrane's Q and quantified by I2. Sources of heterogeneity will be explored by sensitivity and subgroup analyses. A priori subgroup analyses will include nut type, nut dose, duration of follow-up, change in saturated fat intake, change in dietary fibre intake, design (crossover, parallel), study quality, and baseline endpoint values. Significant unexplained heterogeneity will be investigated by additional post hoc subgroup analyses (e.g. age, sex, level of feeding control [metabolic, supplemented, dietary advice], washout in crossover trials, energy balance of the background diet, composition of the background diet [total % energy from fat, carbohydrate, protein], change in cholesterol intake, change in glycemic index, etc.). Meta-regression analyses will assess the significance of subgroups analyses. Publication bias will be investigated by the inspection of funnel plots and application of Egger's and Begg's tests.

Knowledge translation plan: Results from the two systematic reviews and meta-analyses will be disseminated through traditional means such as interactive presentations at local, national, and international scientific meetings and publication in high impact factor journals. Innovative means such as webcasts with e-mail feedback mechanisms will also be used. Knowledge Users will act as knowledge brokers networking among opinion leaders and different adopter groups to increase awareness at each stage. Two of the applicants (JLS, CWCK) will also participate directly as members of nutrition guidelines committees the 2013 CDA Clinical Practice Guidelines (CPG) for nutrition therapy by one of the applicants (JLS) and 2015 European Association for the Study of Diabetes (EASD) CPG for nutrition therapy (JLS, CWCK). Target adopters will include the clinical practice, public health, industry, research communities, and patient groups. Feedback will be incorporated and used to guide analyses and improve key messages at each stage.

Significance: The two proposed systematic reviews and meta-analyses will aid in knowledge translation related to the effects of tree nuts in diabetes and metabolic syndrome, strengthening the evidence-base for dietary recommendations and health claims.

ELIGIBILITY:
Inclusion Criteria:

* Dietary trials in humans
* Randomized treatment allocation
* >=3-weeks
* Suitable control (i.e. isocaloric exchange of other dietary components for tree nuts)
* viable endpoint data

Exclusion Criteria:

* Non-human studies
* Nonrandomized treatment allocation
* 3-weeks
* Lack of a suitable control (non-isocaloric)
* no viable endpoint data

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Varied
Sampling Method: Probability Sample
Enrollment: 1 (Actual)
Dates: Start 2012-05; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Glycemic control measures | Up to 1.5-years
  Glycated blood proteins (HbA1c, total glycated hemoglobin, fructosamine, glycated albumin), fasting glucose, fasting insulin, and the homeostasis model assessment of insulin resistance (HOMA-IR)
Metabolic syndrome measures | Up to 1.5-years
  Harmonized metabolic syndrome diagnostic measures (waist circumference, TG, HDL-C, blood pressure, fasting glucose)

CONTACTS AND LOCATIONS:
Overall Officials: John L Sievenpiper, MD, PhD, Study Director — Department of Pathology and Molecular Medicine, McMaster University and Clinical Nutrition and Risk Factor Modification Centre, St. Michael's Hospital; Russell J de Souza, ScD, RD, Study Director — Department of Epidemiology and Biostatistics, McMaster University and Clinical Nutrition and Risk Factor Modification Centre, St. Michael's Hospital; Cyril WC Kendall, PhD, Principal Investigator — Department of Nutritional Sciences and Medicine, University of Toronto and Clinical Nutrition and Risk Factor Modification Centre, St. Michael's Hospital; David JA Jenkins, MD, PhD, DSc, Principal Investigator — Department of Nutritional Sciences and Medicine, University of Toronto and Clinical Nutrition and Risk Factor Modification Centre, St. Michael's Hospital
Locations (1):
- The Toronto 3D (Diet, Digestive tract and Disease) Knowledge Synthesis and Clinical Trials Unit, Clinical Nutrition and Risk Factor Modification Centre, St. Micheal's Hospital, Toronto, Ontario, Canada

REFERENCES:
- [Background] Jenkins DJ, Kendall CW, Banach MS, Srichaikul K, Vidgen E, Mitchell S, Parker T, Nishi S, Bashyam B, de Souza R, Ireland C, Josse RG. Nuts as a replacement for carbohydrates in the diabetic diet. Diabetes Care. 2011 Aug;34(8):1706-11. doi: 10.2337/dc11-0338. Epub 2011 Jun 29. PMID 21715526 (Retraction: PMID 26798151 Diabetes Care. 2016 Feb;39(2):319)
- [Result] Blanco Mejia S, Kendall CW, Viguiliouk E, Augustin LS, Ha V, Cozma AI, Mirrahimi A, Maroleanu A, Chiavaroli L, Leiter LA, de Souza RJ, Jenkins DJ, Sievenpiper JL. Effect of tree nuts on metabolic syndrome criteria: a systematic review and meta-analysis of randomised controlled trials. BMJ Open. 2014 Jul 29;4(7):e004660. doi: 10.1136/bmjopen-2013-004660. PMID 25074070
- [Result] Viguiliouk E, Kendall CW, Blanco Mejia S, Cozma AI, Ha V, Mirrahimi A, Jayalath VH, Augustin LS, Chiavaroli L, Leiter LA, de Souza RJ, Jenkins DJ, Sievenpiper JL. Effect of tree nuts on glycemic control in diabetes: a systematic review and meta-analysis of randomized controlled dietary trials. PLoS One. 2014 Jul 30;9(7):e103376. doi: 10.1371/journal.pone.0103376. eCollection 2014. PMID 25076495